CLINICAL TRIAL: NCT05339997
Title: Evaluation of Respiratory Function and Functional Capacity in Pediatric Patients With Chronic Kidney Disease (CKD)
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Irmak ÇAVUŞOĞLU, Specialist physiotherapist-Lecturer, Acibadem University
Other Study IDs: ırmak çavuşoğlu
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Diseases; Chronic Renal Disease; Chronic Renal Failure
Keywords: pediatric chronic kidney disease; pulmonary function; functional capacity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 6 minute walk test, — submaximal exercise test used to evaluate the functional capacity of patients
  Other Names: pulmonary function tests

SUMMARY:
Chronic kidney disease (CKD) is defined as a permanent abnormality in kidney structure or function that persists for more than 3 months (for example, glomerular filtration rate [GFR] <60 mL/min/1.73 m2 or albuminuria ≥30 mg/24 hours) and, it effects the 8% to 16% of the population worldwide.In pediatric patients with CKD, exercise capacity begins to decline in stage 3 of the disease and progressively decreases in stage 5, in dialysis and transplant patients (4, 5). Reduction in respiratory muscle strength and six minute walk test (6MWT) is observed in patients with CKD treated with hemodialysis (HD).The aim in present study is to evaluate the relationship between functional capacity and respiratory functions in stage 1-5 pediatric chronic kidney disease patients.

DETAILED DESCRIPTION:
The aim of this study is to evaluate functional capacity with six minutes walk test (6MWT), respiratory functions with spirometer and the correlation between functional capacity and respiratory functions in pediatric CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 5-18, having stage I-V chronic kidney disease,
* Having chronic kidney disease for at least 6 months,
* Not having visual and hearing impairment

Exclusion Criteria:

Presence of mental retardation,

* Insufficient Turkish communication, Inability to communicate,
* Having metabolic-neurological problems,
* Presence of cardiomyopathy, angina pectoris,
* Presence of orthopedic problem that will prevent standing and walking
* Cerebrovascular disease
* Patients will not be included in the study in the presence of metastatic carcinoma.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients aged 5-18 years with stage 1-5 chronic kidney disease
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | during the procedure
  its a submaximal exercise test. The 6MWT is carried out in a marked 30 meter corridor. Patients are asked to walk as quickly as possible. They can stop whenever they want. The distance walked is recorded in meters. And it is interpreted according to the reference values of healthy children.quicly as possible and the distance will be record in meter.

SECONDARY OUTCOMES:
pulmonary function test | during the procedure
  FVC, FEV1, FEV1/FVC, PEF parameters will be eveluated.Patients sit with a clip on their noses. After 3 technically appropriate tests, the best measured values are recorded and compared against reference values.The measurements obtained are recorded as a percentage relative to their ratio to the expected reference values.FEV1, FVC,PEF measurements are recorded as a volume in ml.

CONTACTS AND LOCATIONS:
Overall Officials: Irmak Çavuşoğlu, MSc, Study Director — Acıbadem Mehmet Ali Aydınlar University; Elif Esma Safran, MSc, Study Chair — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Acibadem Mehmet Ali Aydınlar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No